CLINICAL TRIAL: NCT00699010
Title: A Phase II, Single-Center, Randomized, Double-Blind Assessment of the Abuse Liability of Acurox (Oxycodone HCl and Niacin) Tablets in Subjects With a History of Opioid Abuse
Brief Title: Study of the Abuse Liability of Oxycodone HCl/Niacin in Subjects With a History of Opioid Abuse
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Acura Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AP-ADF-111
Record Dates: First submitted 2008-06-13; First posted 2008-06-17 (Estimated); Results first posted 2018-10-03 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2008-10

CONDITIONS: Opioid Abuse
Keywords: Abuse Liability; Abuse Prevention; Abuse Resistance; Abuse Deterrence
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Oxycodone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acurox 5/30mg taken first (Active Comparator): oxycodone HCl/Niacin 5/30mg tablets; 8 tablets per dose
  Interventions: Drug: Acurox 5/30mg taken first
- Oxycodone 5mg taken first (Active Comparator): oxycodone HCl 5mg tablets; 8 tablets per dose
  Interventions: Drug: Oxycodone 5mg taken first

INTERVENTIONS:
Drug: Acurox 5/30mg taken first — followed by oxycodone 5mg with 48 hour washout
  Arms: Acurox 5/30mg taken first
Drug: Oxycodone 5mg taken first — followed by Acurox 5/30mg with 48 hour washout
  Arms: Oxycodone 5mg taken first

SUMMARY:
The purpose of this study is to assess the abuse liability of 4 times (8 tablets) the usual recommended dose of Acurox (oxycodone HCl 40 mg plus niacin 240 mg) versus oxycodone HCL 40 mg alone in subjects with a history of opioid abuse.

DETAILED DESCRIPTION:
In the Treatment Phase, subjects randomly received oxycodone HCl 40 mg administered in combination with niacin 240 mg and oxycodone HCl 40 mg alone in crossover design. 15 subjects were randomized to receive oxycodone/niacin first followed by oxycodone with a 48 hour washout between doses. 15 subjects randomized to receive oxycodone before the oxycodone/naicin dose with a 48 hour washout between doses. The purpose of the Treatment Phase was to assess the abuse liability and abuse deterrence potential of 4 times the recommended 2-tablet dose of Acurox® Tablets 5/30 mg versus oxycodone HCl 40 mg alone (8 tablets per dose).

All 30 subjects received a single dose of each study treatment. Subjects were fasted prior to dosing on all dose days.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female between 18 and 55 years of age
* Subject meets DSM-IV Criteria for the Diagnosis of Opioid Substance Abuse and subject is unlikely to experience an idiosyncratic reaction or respiratory depression after ingesting 40 mg of oxycodone
* Body weight is not more than 20% above or below ideal body weight
* Subject agrees to abstain from any Rx or OTC drugs (except as authorized by the Investigator) or alcohol
* Subject is in generally good health
* Subject is reliable, willing, cooperative, able to communicate effectively, and has a minimum of a 6th grade reading level
* Subject has an acceptable score on the MMSE for cognitive impairment
* For women of child-bearing potential: woman is not pregnant and not nursing, and is practicing an acceptable method of birth control

Exclusion Criteria:

* Subject has a disease that may endanger the subject or the validity of the data
* Subject is currently physically dependent on opiates or alcohol
* Subject was exposed to any investigational drug within 30 days prior to the inpatient phase
* Subject has a history of hypersensitivity to any drug, or a known allergy to any component of the study drug formulation
* Subject has a positive urine drug screen for a non-opiate drug
* Subject has a predisposing condition that may place the subject at risk for receiving niacin or oxycodone, or confound the study analyses
* Subject ingested niacin at doses higher than SDI within 14 days prior to the inpatient phase
* Subject has an abnormal bleeding tendency

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2008-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald R Jasinski, MD, Principal Investigator — Johns Hopkins Medical Center
Locations (1):
- Johns Hopkins Medical Center, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Acurox 5/30mg Taken First: Oxycodone HCl/Niacin 5/30mg; 8 tablet dose followed by oxycodone 5mg with 48 hour washout
- Oxycodone 5mg Taken First: Oxycodone Hcl 5mg; 8 tablet dose follwed by Acurox 5/30mg with 48 hour washout
Period: Overall Study
Arm/Group | Acurox 5/30mg Taken First | Oxycodone 5mg Taken First
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Recreational Drug Abusers
Groups:
- Oxycodone 5mg Taken First: Oxycodone HCL 5mg; 8 tablet dose followed by Acurox 5/30mg with 48 hour washout
- Total: Total of all reporting groups
Arm/Group | Acurox 5/30mg Taken First | Oxycodone 5mg Taken First | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.7 (5.5) | 44.7 (5.5) | 44.7 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 13 | 13 | 26
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 39

OUTCOME MEASURES:

1. Primary Outcome: Drug Like/Dislike Effect at 30 Minutes Post Dose (E 30 Min)
Description: "Do you dislike or like the drug effect you are feeling now?" This question was rated on a 1 to 29 point VAS scale that was anchored in the center with "neither like nor dislike" (14), on the left with "dislike an awful lot" (1), and on the right with "like an awful lot" (29).
Time Frame: Effects assessed at 0.5 hours after dosing.
Population: Study completers and per protocol
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Acurox 5/30mg: Oxycodone HCL/Niacin 5/30mg; 8 tablet dose
- Oxycodone 5mg: Oxycodone 5mg; 8 tablet dose
Arm/Group | Acurox 5/30mg | Oxycodone 5mg
Number analyzed (Participants) | 30 | 30
score on a scale | 11.7 (1.0) | 14.7 (1.0)

ADVERSE EVENTS:
Time Frame: 11 days. Doses taken 1 per day with a 48 hours washout
Groups:
- Oxycodone 5mg: Oxycodone HCl 5mg; 8 tablet dose
Arm/Group | Acurox 5/30mg | Oxycodone 5mg
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 28/30 | 29/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acurox 5/30mg (N=30) | Oxycodone 5mg (N=30)
Flushing (Vascular disorders) | 23 (23) | 5 (5) — Flushing
Pruritis (Skin and subcutaneous tissue disorders) | 21 (21) | 21 (21)
Nausea (Gastrointestinal disorders) | 8 (8) | 9 (9)
Euphoria (Nervous system disorders) | 13 (13) | 15 (15)
Paraesthesia (Skin and subcutaneous tissue disorders) | 11 (11) | 3 (3)
Somnolence (Nervous system disorders) | 8 (8) | 9 (9)
Vomiting (Gastrointestinal disorders) | 4 (4) | 3 (3)
Headache (Nervous system disorders) | 8 (8) | 7 (7)
Dizziness (Nervous system disorders) | 6 (6) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No